CLINICAL TRIAL: NCT02552966
Title: Assessing the Impacts of an Upper Esophageal Sphincter Assist Device on Laryngeal Symptoms and Salivary Pepsin: A Pilot Study
Brief Title: Assessing the Impacts of a UESAD on Laryngeal Symptoms and Salivary Pepsin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Somna Therapeutics, L.L.C. (Industry)
Responsible Party: Principal Investigator, John Pandolfino, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00201370
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-07

CONDITIONS: Laryngopharyngeal Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UESAD (Experimental): Upper Esophageal Sphincter Assist Device
  Interventions: Device: UESAD

INTERVENTIONS:
Device: UESAD — Device designed to provide modest cricoid pressure to reduce reflux

SUMMARY:
It is postulated that the incompetence of the upper esophageal sphincter (UES) to restrict passage of esophageal refluxate is fundamental to the development of LPR. The UES Assist Device (UESAD) is a novel device that applies relatively modest external cricoid pressure, which results in a 20 to 30 mmHg intraluminal UES pressure increase. Pepsin, a proteolytic enzyme produced in the stomach, has been detected in the laryngeal epithelium of patients with reflux associated laryngeal symptoms and implicated in the pathogenesis of laryngopharyngeal reflux. This study will assess the effectiveness of a UESAD worn for 2 weeks on LPR symptoms and salivary pepsin levels.

DETAILED DESCRIPTION:
A cost-effective and care appropriate algorithm to streamline the diagnosis and management of patients with laryngopharyngeal reflux (LPR) has not been described. It is postulated that the incompetence of the upper esophageal sphincter (UES) to restrict passage of esophageal refluxate is fundamental to the development of LPR. The UES Assist Device (UESAD) is a novel device that applies relatively modest external cricoid pressure, which results in a 20 to 30 mmHg intraluminal UES pressure increase. Pepsin, a proteolytic enzyme produced in the stomach, has been detected in the laryngeal epithelium of patients with reflux associated laryngeal symptoms and implicated in the pathogenesis of laryngopharyngeal reflux. A study examining salivary pepsin levels for patients pre- and post-fundoplication for LPR found that all patients with positive preoperative pepsin levels and postoperative elimination had symptom improvement, suggesting that changes in pepsin level may be reflective of surgical responsiveness. This study seeks to explore the therapeutic role of the UESAD in patients with LPR symptoms, and measure its effectiveness by objective criteria (salivary pepsin) and symptomatic improvement. In this study, 25 patients seen in GI clinic with laryngeal complaints will complete validated symptom questionnaires - the RSI, GerdQ and N-GSSIQ scores. Those with an RSI > 13 and GerdQ > 8 will be included. They will submit 3 baseline sputum samples for pepsin analysis, taken upon awaking. They will then be advised to use the UESAD nightly for 2 weeks. 3 follow-up sputum samples for pepsin analysis will be taken and symptom scores reevaluated after the 2 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female persons age 18-90
2. Patients with LPR symptoms (RSI >13)

Exclusion Criteria:

1. Pregnant patients per history on initial evaluation.
2. Adults unable to consent in English
3. Patients who are currently imprisoned
4. Patients started on PPI therapy within 4 weeks of study
5. Patients with implants or implant parts that reside in the area where the REZA BAND is applied.
6. Patients with an implanted pacemaker, implanted cardioverter defibrillator (ICD), vagus nerve stimulator, or other such similar devices implanted in the neck.
7. Patients diagnosed with glaucoma.
8. Patients who had a malignancy of the neck, including neck surgery.
9. Patients that may have an altered mental status including due to the use of sedative drugs or narcotics.
10. Patients with carotid artery disease, thyroid disease, a history of cerebrovascular disease, or any disorder of connective tissues (e.g., Marfan's Syndrome or Ehlers-Danlos Syndrome).
11. Patients who use nocturnal NIV machines such as CPAP or BiPAP.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Pandolfino, MD, Principal Investigator — Northwestern University

REFERENCES:
- [Background] El-Serag HB, Lee P, Buchner A, Inadomi JM, Gavin M, McCarthy DM. Lansoprazole treatment of patients with chronic idiopathic laryngitis: a placebo-controlled trial. Am J Gastroenterol. 2001 Apr;96(4):979-83. doi: 10.1111/j.1572-0241.2001.03681.x. PMID 11316215
- [Background] Francis DO, Rymer JA, Slaughter JC, Choksi Y, Jiramongkolchai P, Ogbeide E, Tran C, Goutte M, Garrett CG, Hagaman D, Vaezi MF. High economic burden of caring for patients with suspected extraesophageal reflux. Am J Gastroenterol. 2013 Jun;108(6):905-11. doi: 10.1038/ajg.2013.69. Epub 2013 Apr 2. PMID 23545710
- [Derived] Yadlapati R, Craft J, Adkins CJ, Pandolfino JE. The Upper Esophageal Sphincter Assist Device Is Associated With Symptom Response in Reflux-Associated Laryngeal Symptoms. Clin Gastroenterol Hepatol. 2018 Oct;16(10):1670-1672. doi: 10.1016/j.cgh.2018.01.031. Epub 2018 Jan 31. PMID 29408585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Northwestern Medicine Gastroenterology clinic during the study period beginning 9/1/2015. A total of 15 subjects
Period: Overall Study
Arm/Group | UESAD
Started | 20
Completed | 15
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | UESAD
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 45.7 [27 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
GERDQ [Mean (Standard Deviation); unit: units on a scale] — GastroEsophageal Reflux Disease Questionnaire (GERDQ). This scale measures symptom burden of gastroesophageal reflux disease (GERD). A higher score indicated greater symptom severity on a scale of 0 to 18. No subscales are combined to compute the total score. "Units on a scale" is the appropriate Unit of Measure.
  units on a scale | 10.4 (2.1)
Reflux Symptom Index (RSI) [Mean (Standard Deviation); unit: units on a scale] — Reflux Symptom Index (RSI). This questionnaire measures laryngeal symptom severity for subjects experiencing reflux-related laryngeal symptoms (e.g. sore throat, throat clearing, post nasal drip, globus and cough). A higher score indicates greater severity on a scale of 0 to 45. No subscales are used to compute a total score. "Units on a scale" is the appropriate unit of measure for this questionnaire.
  units on a scale | 26.0 (7.8)
NGSSIQ [Mean (Standard Deviation); unit: units on a scale] — Nocturnal GERD Symptom Severity & Impact Questionnaire (NGSSIQ). This questionnaire assesses nighttime symptom severity and the impact of nighttime GERD symptoms. A higher scoe indicates greater severity on a scale of 0 to 60. No subscales were used to calculate the composite score. "Units on a scale" is the appropriate unit of measure for this questionnaire.
  units on a scale | 43.4 (20.1)
Pepsin (ng/mL) [Mean (Standard Deviation); unit: ng/mL] — Salivary Pepsin (referred to as "pepsin") is a biomarker measured in this study in ng/mL.
  ng/mL | 146.5 (172.7)

OUTCOME MEASURES:

1. Primary Outcome: Salivary Pepsin Concentration
Description: Average salivary pepsin concentration
Time Frame: 2 weeks
Population: Twelve subjects provided post-treatment salivary samples for pepsin analysis. While the subject flow shows 20 subjects (all of which completed baseline pepsin analysis), only 12 completed post-treatment testing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | UESAD
Number analyzed (Participants) | 12
ng/mL | 158.4 (150.2)
Statistical Analysis 1: Comparison: UESAD; Test type: Other; p = 0.61, t-test, 2 sided; This t-test was applied to determine if the mean salivary pepsin concentration changed between baseline and 2 week post UESAD measurements

2. Secondary Outcome: RSI Score
Description: Respiratory symptom index (RSI) score. Values between 0 and 45. Higher value is associated with increased symptom severity.
Time Frame: 2 weeks
Population: 15 subjects completed the RSI post-treatment. The subject flow shows 20 subjects completing this questionnaire at baseline, but this section reflects the 15 subjects who completed this questionnaire post-treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UESAD
Number analyzed (Participants) | 15
units on a scale | 19.4 (8.5)
Statistical Analysis 1: Comparison: UESAD; Test type: Other; p < 0.01, t-test, 2 sided

3. Secondary Outcome: GerdQ Score
Description: GERDQ score. Scale of 0-12, higher score indicates increased symptom severity.
Time Frame: 2 weeks
Population: Fifteen subjects completed the post-treatment GERDQ questionnaire. While 20 subjects completed the questionnaire at baseline, this section contains results from the 15 who completed the questionnaire 2 weeks post UESAD treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UESAD
Number analyzed (Participants) | 15
units on a scale | 8.6 (2.4)
Statistical Analysis 1: Comparison: UESAD; Test type: Other; p < 0.01, t-test, 2 sided

4. Secondary Outcome: NGSSIQ Score
Description: NGSSI questionnaire score
Time Frame: 2 weeks
Population: Fifteen subjects completed the post-treatment questionnaire. While 20 subjects (as indicated on the participant flow section) completed the baseline questionnaire, this section reflects the results of the 15 subjects who completed the questionnaire at 2 weeks post UESAD treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UESAD
Number analyzed (Participants) | 15
units on a scale | 26.8 (20.8)
Statistical Analysis 1: Comparison: UESAD; Test type: Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 days
Description: adverse events were collected throughout the study
Arm/Group | UESAD
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02552966/Prot_SAP_000.pdf